CLINICAL TRIAL: NCT05701904
Title: Investigation of the Effect of Local Mechanical Vibration and Shotblocker Application on Pain and Patient Satisfaction Before Tetanus + Diphtheria Vaccine in Pregnant Women
Brief Title: Vibration and Shotblocker Use in Pregnant Women While Giving Tetanus + Diphtheria Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Senem Andı, RN, Doktora Öğrencisi, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HKU-SBF-SA-01
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pain
Keywords: Nursing care; Management, Pain; Patient Satisfaction; Intramuscular Injections
MeSH Terms: conditions — Pain; Agnosia; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: a control group and 2 intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local mechanical vibration applied group (Experimental): Before the injection, local mechanical vibration will be applied for 3 minutes with a vibration device to the deltoid muscle where the injection will be made, and then the vaccine will be given. The vibration device to be used is suitable for contact with the skin and provides 6000 rotations per minute with vibration.
  Pregnant women who were asked to receive tetanus+diphtheria vaccine by their physician and agreed to participate in the study will be informed about the research by the researcher, and their written and verbal consents will be obtained. Then the vaccine will be administered. Td vaccine will be administered to all pregnant women in the study as IM to the deltoid muscle in the arm they do not use dominantly. Five minutes after the vaccination, the individual descriptor form will be applied to all pregnant women, and the pregnant women will score their satisfaction levels with regard to pain and the method used.
  Interventions: Other: Local mechanical vibration
- Shotblocker group (Experimental): It is a U-shaped device with skin contact points on the shotblocker and an opening in the middle for injecting. The Shotblocker will be placed on the skin surface just before inserting the needle and gently pressed with the fingertips, and the vaccine will be administered immediately afterwards. After removing the needle, the shotblocker will be removed.
  Pregnant women who were asked to receive tetanus+diphtheria vaccine by their physician and agreed to participate in the study will be informed about the research by the researcher, and their written and verbal consents will be obtained. Then the vaccine will be administered. Td vaccine will be administered to all pregnant women in the study as IM to the deltoid muscle in the arm they do not use dominantly. Five minutes after the vaccination, the individual descriptor form will be applied to all pregnant women, and the pregnant women will score their satisfaction levels with regard to pain and the method used.
  Interventions: Other: Shotblocker group
- Control group (No Intervention): The vaccine will be administered by following the standard intramuscular injection procedure. Five minutes after vaccination, an individual descriptive form will be applied to all pregnant women, and pregnant women will score their pain and satisfaction levels with scales.
  Pregnant women who were asked to receive tetanus+diphtheria vaccine by their physician and agreed to participate in the study will be informed about the research by the researcher, and their written and verbal consents will be obtained. Then the vaccine will be administered. Td vaccine will be administered to all pregnant women in the study as IM to the deltoid muscle in the arm they do not use dominantly. Five minutes after the vaccination, the individual descriptor form will be applied to all pregnant women, and the pregnant women will score their satisfaction levels with regard to pain and the method used.

INTERVENTIONS:
Other: Local mechanical vibration — Before the injection, local mechanical vibration will be applied for 3 minutes with a vibration device to the deltoid muscle where the injection will be made, and then the vaccine will be given. The vibration device to be used is suitable for contact with the skin and provides 6000 rotations per minute with vibration.
  Arms: Local mechanical vibration applied group
Other: Shotblocker group — It is a U-shaped device with skin contact points on the shotblocker and an opening in the middle for injection (Tugrul, Celik, and Khorshid 2017). The Shotblocker will be placed on the skin surface just before inserting the needle and gently pressed with the fingertips, and the vaccine will be administered immediately afterwards. After removing the needle, the shotblocker will be removed.
  Arms: Shotblocker group

SUMMARY:
Tetanus-diphtheria vaccine administered to pregnant women may cause pain during and after administration. Due to the pain that may occur, the compliance of pregnant women towards the vaccine may be impaired. Therefore, there is a need for methods that are safe for pregnant women to reduce pain. One of the applications used to reduce pain during intramuscular injection is local mechanical vibration application. With the application of vibration, the tactile receptors are stimulated and the pain is localized in a more limited area. One of the methods used to reduce the pain felt during intramuscular injection is the application of shotblocker applied to the injection site. The protrusions on the Shotbloker temporarily suppress the pain thanks to the pressure it exerts on the skin. Thus, the gates to the central nervous system are closed and pain is reduced. Mechanical vibration and shotblocker procedures applied before injection are non-invasive. Being simple and safe, it is one of the appropriate methods that can be preferred by pregnant women to reduce injection pain. Therefore, in our study, it is aimed to examine the effect of local mechanical vibration and shotblocker application on pain and patient satisfaction before tetenosis-diphtheria vaccine in pregnant women.

DETAILED DESCRIPTION:
Pregnant women who meet the inclusion criteria of the study, who request tetanus-diphtheria (0.5 ml) by their family physician, and who agree to participate in the study will be informed about the study and their written and verbal consents will be obtained. Then the vaccine will be administered. Tetanus-diphtheria vaccine will be administered to all pregnant women in the study by IM in the deltoid muscle in the arm they do not use dominantly.

Data Collection Tools Individual Introduction Form It was prepared by the researchers by scanning the literature . In the introductory form, there are questions about the age, education level, marital status, occupation, income status, smoking status, gestational week, tetonosis vaccination status, height-weight of the pregnant women.

Visual Analog Scale (VAS) VAS patients are initially painless and eventually represent the most severe pain they can feel.

It is a 100 mm straight horizontal line with numbers 0 to 10. '0' means no pain, '10' means severe pain. Participants are asked to mark any number between "0" and "10".

Visual Patient Satisfaction Scale Visual patient satisfaction scale (visual analogue patient satisfaction scale) overlaps with the features of VAS. It indicates the degree of satisfaction out of 10. On one side of the scale, "0" (Not at all satisfied) and on the other side "10" (Very satisfied).

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteered to participate in the study and received written consent
* Pregnant women who were prescribed tetanus + diphtheria vaccine
* No acute cause of pain other than injection pain
* Able to communicate verbally
* Pregnant women over the age of 18

Exclusion Criteria:

* Not willing to participate in the study
* Pregnant women who are not prescribed tetanus + diphtheria vaccine
* An acute cause of pain other than injection pain
* Unable to communicate verbally
* Pregnant women under the age of 18
* Those over the age of 18 who are not pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women with tetanus + diphtheria vaccination order
Enrollment: 96 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 months
  The VAS is a 100 mm straight horizontal line with numbers from 0 to 10 representing the patient's initial pain-free and finally the most severe pain they can feel. '0' means no pain, '10' means severe pain. Participants are asked to mark any number between "0" and "10".

SECONDARY OUTCOMES:
Visual Patient Satisfaction Scale | 4 months
  Visual patient satisfaction scale (visual analog patient satisfaction scale) overlaps with the features of the Visual Analog Scale. It indicates the degree of satisfaction out of 10. On one side of the scale, "0" (Not at all satisfied) and "10" (Very satisfied) are on the other side.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Dincer B, Yildirim D. The effect of vibration stimulation on intramuscular injection pain and patient satisfaction: Single-blind, randomised controlled study. J Clin Nurs. 2021 Jun;30(11-12):1615-1622. doi: 10.1111/jocn.15715. Epub 2021 Mar 1. PMID 33590594